CLINICAL TRIAL: NCT06076486
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Trial to Evaluate the Efficacy and Safety of Elagolix Tablets in Patients With Moderate or Severe Endometriosis-associated Pain
Brief Title: A Clinical Trial to Evaluate Efficacy and Safety of Elagolix Tablets in Women With Moderate or Severe Endometriosis-associated Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALGKNP2022-III
Record Dates: First submitted 2023-09-13; First posted 2023-10-10 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elagolix 200 mg BID (Experimental): Participants received elagolix 200 mg tablets twice a day (BID)
  Interventions: Drug: Elagolix
- Elagolix placebo (Placebo Comparator): Participants received elagolix placebo twice a day (BID)
  Interventions: Drug: Elagolix placebo

INTERVENTIONS:
Drug: Elagolix — Elagolix 200 mg tablets administered orally BID
  Arms: Elagolix 200 mg BID
Drug: Elagolix placebo — Elagolix placebo administered orally BID
  Arms: Elagolix placebo

SUMMARY:
This is a phase 3, multicenter, double-blind, placebo-controlled, randomized study to evaluate the efficacy and safety of elagolix tablets versus placebo in premenopausal women with moderate or severe endometriosis-associated pain.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and methods, voluntarily participate in this trial, and sign the informed consent.
2. Diagnosis of endometriosis by pathological diagnosis or surgery within 10 years prior to screening by laparoscopy or exploratory laparotomy; or diagnosis of endometriosis based on clinical presentation of endometriosis in combination with previous imaging studies according to Endometriosis Diagnosis and Treatment Guidelines (Third Edition).
3. Premenopausal female aged 18 and 49 years (both inclusive) with one complete menstruation prior to screening record in the diary for at least 35 days and at least one complete menstrual cycle before the first dosing.
4. Agree to take only protocol-specified permitted rescue analgesic medications during the screening and treatment Periods.
5. Cervical smear is normal or abnormal without clinical significance (acceptance of normal cervical smear within 6 months prior to screening; or participant is virgin and decides not to take cervical smear); ASCUS may be combined with HPV testing. ASCUS participants may be included if they are negative for high-risk HPV.
6. Agree to use non-hormonal contraception from signing the informed consent through 1 month after last dosing.

Exclusion Criteria:

1. Subjects with a history of sensitivity to elagolix or excipients; or with a known history of serious, life-threatening or significant allergy to any drug.
2. Previous non-responders to GnRH agonist or GnRH antagonist therapy as judged by the investigator.
3. Subjects with a history of previous or existing osteoporosis or other metabolic bone disease; or previous abnormal clinically significant hypocalcemia, hypophosphatemia or hyperphosphatemia; or DXA Z score (subjects < 40 years old) or T score (subjects ≥ 40 years old) of lumbar spine (L1-L4), femoral neck or total hip BMD is < -2.0;
4. Subjects with unstable diseases (such as poorly controlled diabetes, poorly controlled hypertension, poorly controlled seizures, unstable angina pectoris, inflammatory bowel disease, hyperprolactinemia, malignant tumors (except basal cell carcinoma of the skin) or severe infection, etc.) unuitable for the study at screening as judged by the investigators;
5. Subjects with a history of hysterectomy, oophorectomy, or surgery affecting drug absorption; or those who plan to undergo the above surgery during the trial;
6. Subjects with a history of major depressive disorder or post-traumatic stress disorder within 2 years prior to screening or other major psychiatric disorder at any time (e.g., schizophrenia, bipolar disorder); or history of suicidal behavior or suicidality; or suicidality as judged by the investigators;
7. Subjects with undiagnosed vaginal and/or uterine bleeding within 3 months prior to screening;
8. Subjects with other chronic pain syndromes requiring chronic analgesia or other long-term treatment that would be expected to interfere with the assessment of endometriosis-related pain;
9. Subjects with a history of drug or alcohol abuse within 6 months prior to screening;
10. Subjects aged ≥ 40 years with abnormal results of breast ultrasonography during the screening period or within 1 year prior to screening (BI-RADS classification grade 4 and above);
11. Clinically significant gynecological conditions (e.g., any non-malignant cyst > 6 cm, or malignant cyst) by TVU or transrectal ultrasound or transabdominal ultrasound at screening;
12. Subjects with hepatitis B [HbsAg is positive and detection of HBV-DNA indicates viral replication], hepatitis C [HCV antibody is positive and detection of HCV-RNA indicates viral replication], positive syphilis (except specific antibody detection positive, non-specific antibody detection negative and confirmed as inactive infection in combination with clinical judgment), known HIV positive history or HIV positive;
13. Subjects with moderate/severe liver injury caused by previous diseases, or AST or ALT or bilirubin ≥ 2 × ULN at screening;
14. Subjects requiring the use of a prohibited long-acting anesthetic or immediate-release anesthetic for more than 2 consecutive weeks for the treatment of endometriosis-related pain within 6 months prior to screening;
15. Participation in any other interventional clinical trial (including drug and device clinical trials) within 1 month prior to screening;
16. Use of any systemic corticosteroids for more than 2 weeks within 3 months prior to screening or likely to require such therapy during the study (topical, inhaled, or nasal corticosteroids are allowed);
17. Use of GnRH agonists or GnRH antagonists (including participation in clinical trails of elagolix) within 6 months prior to screening; use of medroxyprogesterone acetate, danazol, aromatase inhibitors within 3 months prior to screening; use of oral contraceptives, or any hormonal treatment for endometriosis within 2 months prior to screening; use of Chinese herbal medicine for endometriosis treatment or symptom relief within 1 month prior to screening;
18. Subjects with IUD or subcutaneous contraceptive implants (the IUD or subcutaneous contraceptive implants removed more than 30 days prior to screening is allowed);
19. Subjects taking moderate or strong CYP450 3A inducers or OATP1B1 inhibitors within 1 month prior to the first dosing;
20. Pregnant or lactating women; or plan to have children during the trial (from signing the informed consent form to 3 months after using the study drug); or < 6 months after delivery; or < 3 months after abortion; or have a positive pregnancy test result during the screening period or on the day of randomization;
21. Subjects with increasing risk associated with the study, interference with the interpretation of study results, or inappropriate as judged by the investigators.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 202 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Percentage of responders of dysmenorrhea (DYS) at week 12 | 12 weeks
  The responder was defined as reaching a pre-defined threshold.
Percentage of responders of Non-Menstrual Pelvic Pain (NMPP) at week 12 | 12 weeks
  The responder was defined as reaching a pre-defined threshold.

SECONDARY OUTCOMES:
Change from baseline in DYS | Through study completion, an average of 24 weeks
  The DYS pain scale s range from 0 (none) to 3 (severe).
Change from baseline in NMPP | Through study completion, an average of 24 weeks
  The NMPP pain scales range from 0 (none) to 3 (severe).
Change from baseline in Dyspareunia (DYSP) | Through study completion, an average of 24 weeks
  The DYSP pain scales range from 0 (none) to 3 (severe).
Change from baseline in Numeric Rating Scale (NRS) scores | Through study completion, an average of 24 weeks
  The NRS pain scores ranges 0 (none) to 10 (worst pain ever).
Change from baseline in rescue analgesic use | Through study completion, an average of 24 weeks
  Use of rescue analgesic medications taken for endometriosis-associated pain was recorded by the subject daily as the total number of pills/tablets of each type taken within a 24-hour period.
Percentage of participants with a Patient Global Impression of Change (PGIC) response | Through study completion, an average of 24 weeks
  PGIC response was defined as very much improved and much improved selected by the subject to assess the change in endometriosis-associated pain since the initiation of study drug.
Safety Specifications in the Treatment Period | Through study completion, an average of 24 weeks
  AEs and SAEs occurred during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfang Zhou, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No